CLINICAL TRIAL: NCT00178022
Title: A Trial of Two On-Line Interventions for Child Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: 0410002
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Traumatic Brain Injury; Depression; Anxiety Disorders
Keywords: tbi; intervention; depression; anxiety
MeSH Terms: conditions — Brain Injuries, Traumatic; Depression; Anxiety Disorders | interventions — Case Management

INTERVENTIONS:
Behavioral: Case management and problem solving therapy

SUMMARY:
The primary aims of this project are to examine the feasibility and relative efficacy of two models of on-line intervention for families of children with traumatic brain injury: one, a model emphasizing cognitive appraisals and problem solving skills; the other, emphasizing linking families to resources and providing professionally-moderated peer support.

DETAILED DESCRIPTION:
The feasibility of the two interventions will be evaluated by examining family utilization of on-line materials and satisfaction with receiving services this way. Previous studies suggest the longer-term effects of TBI often create significant stress for both child and family and the need for psychological services.

ELIGIBILITY:
Inclusion Criteria:

* Child between 5 and 17 years old who experienced a TBI in the past 12 months

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120
Dates: Start 2005-02; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Previous investigations using problem solving therapy have documented large effect sizes on measures of problem solving and depression.

SECONDARY OUTCOMES:
Similarly, the single previous controlled intervention following pediatric traumatic brain injury (TBI) demonstrated a large effect on self-report measures of depression and anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Armando J Rotondi, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Wade SL, Fisher AP, Kaizar EE, Yeates KO, Taylor HG, Zhang N. Recovery Trajectories of Child and Family Outcomes Following Online Family Problem-Solving Therapy for Children and Adolescents after Traumatic Brain Injury. J Int Neuropsychol Soc. 2019 Oct;25(9):941-949. doi: 10.1017/S1355617719000778. Epub 2019 Aug 13. PMID 31405391
- [Derived] Wade SL, Kaizar EE, Narad M, Zang H, Kurowski BG, Yeates KO, Taylor HG, Zhang N. Online Family Problem-solving Treatment for Pediatric Traumatic Brain Injury. Pediatrics. 2018 Dec;142(6):e20180422. doi: 10.1542/peds.2018-0422. Epub 2018 Nov 9. PMID 30413559